CLINICAL TRIAL: NCT03356821
Title: Adult Mesenchymal Stromal Cells to Regenerate the Neonatal Brain: the PASSIoN Trial (Perinatal Arterial Stroke Treated With Stromal Cells IntraNasally)
Brief Title: Perinatal Arterial Stroke Treated With Stromal Cells Intranasally
Acronym: PASSIoN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, dr. M.J.N.L. Benders, MD, PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL59265.000.16
Record Dates: First submitted 2017-11-08; First posted 2017-11-29 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-12

CONDITIONS: Perinatal Arterial Ischemic Stroke; Neonatal Stroke

STUDY DESIGN:
Intervention Model Description: A phase I/II, open-label, single-arm, single-center intervention study in the NICU at the Wilhelmina children's Hospital / University Medical Centre in Utrecht of (near-)term newborns ≥36 weeks of gestation within the first week of onset of presenting clinical symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cells (Experimental): All (near-)term newborns ≥36 weeks of gestation with or without clinical symptoms of PAIS but with a magnetic resonance imaging (MRI) confirmed PAIS (in the Middle Cerebral Artery region) will be eligible for this study. Following written parental consent, 10 patients will be included in our study.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — One dose of 50x10^6 bone marrow-derived allogeneic MSCs via the nasal route as soon as possible after confirmation of the stroke (in the middle cerebral artery), but within the first week of onset of presenting clinical symptoms. Within 30 minutes after cleaning the nose with saline, using standard procedures operative at the Neonatal Intensive Care Unit, the MSC will be delivered.
  Other Names: Bone Marrow-derived Allogeneic Mesenchymal Cells

SUMMARY:
This study will assess safety and feasibility of bone marrow-derived allogeneic MSCs, administered by the nasal route, in neonates who suffered from PAIS.

DETAILED DESCRIPTION:
Perinatal arterial ischemic stroke (PAIS) is an important perinatal cause of long-lasting neurodevelopmental problems. Recent studies report an incidence of PAIS of 1 per 2300 full-term infants born alive. Adverse consequences of PAIS include hemiplegia, cognitive dysfunction, epilepsy and speech problems. In 50-75% of infants, neonatal stroke leads to abnormal neuromotor and -developmental outcome or epilepsy. The estimated annual mortality rate of neonatal stroke is 3.49/100,000 annually. Current treatment options for PAIS mainly focus on controlling convulsions and associated infections. There is no treatment available that leads to reduction of neonatal brain damage in this severely affected group of infants. This leads to life-long consequences of PAIS and forms a large burden for patients and society. The overall aim of this project is to meet this need by developing a cell based treatment strategy. Animal models of neonatal brain injury provide evidence for the feasibility and efficacy of intranasal mesenchymal stromal cell (MSC) application in the treatment of PAIS. Additionally, results from human trials with MSCs in the treatment of adult stroke or other pathologic conditions provide evidence that MSC treatment is safe. This project aims at making the first step towards clinical application of MSCs to treat PAIS. Successful completion of this project will provide the first evidence of the safety and feasibility of MSCs to treat brain damage in newborn infants. This study will assess safety and feasibility of bone marrow-derived allogeneic MSCs, administered by the nasal route, in neonates who suffered from PAIS.

ELIGIBILITY:
Inclusion Criteria:

* (Near-)Term infants, ≥36+0 weeks of gestation, admitted to one of the Dutch Neonatal Intensive Care Units, diagnosed with PAIS, confirmed by MRI within 3 days after presentation with clinical symptoms.
* PAIS as characterized by a predominantly unilateral ischemic lesion within the territory of the middle cerebral artery, with involvement of the corticospinal tracts, cortex, white matter and basal ganglia.
* Written informed consent from custodial parent(s).

Exclusion Criteria:

* Any proven or suspected congenital anomaly, chromosomal disorder, metabolic disorder.
* Presence of an infection of the central nervous system.
* No realistic prospect of survival, (e.g. severe brain injury), at the discretion of the attending physician.

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manon Benders, MD, PhD, Principal Investigator — UMC Utrecht; Floris Groenendaal, MD, PhD, Principal Investigator — UMC Utrecht; Frank van Bel, MD, PhD, Principal Investigator — UMC Utrecht; Cora Nijboer, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- Wilhelmina Childrens Hostpital/University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Donega V, van Velthoven CT, Nijboer CH, Kavelaars A, Heijnen CJ. The endogenous regenerative capacity of the damaged newborn brain: boosting neurogenesis with mesenchymal stem cell treatment. J Cereb Blood Flow Metab. 2013 May;33(5):625-34. doi: 10.1038/jcbfm.2013.3. Epub 2013 Feb 13. PMID 23403379
- [Background] Donega V, van Velthoven CT, Nijboer CH, van Bel F, Kas MJ, Kavelaars A, Heijnen CJ. Intranasal mesenchymal stem cell treatment for neonatal brain damage: long-term cognitive and sensorimotor improvement. PLoS One. 2013;8(1):e51253. doi: 10.1371/journal.pone.0051253. Epub 2013 Jan 3. PMID 23300948
- [Background] Donega V, Nijboer CH, van Tilborg G, Dijkhuizen RM, Kavelaars A, Heijnen CJ. Intranasally administered mesenchymal stem cells promote a regenerative niche for repair of neonatal ischemic brain injury. Exp Neurol. 2014 Nov;261:53-64. doi: 10.1016/j.expneurol.2014.06.009. Epub 2014 Jun 16. PMID 24945601
- [Background] Donega V, Nijboer CH, Braccioli L, Slaper-Cortenbach I, Kavelaars A, van Bel F, Heijnen CJ. Intranasal administration of human MSC for ischemic brain injury in the mouse: in vitro and in vivo neuroregenerative functions. PLoS One. 2014 Nov 14;9(11):e112339. doi: 10.1371/journal.pone.0112339. eCollection 2014. PMID 25396420
- [Background] van Velthoven CT, Kavelaars A, Heijnen CJ. Mesenchymal stem cells as a treatment for neonatal ischemic brain damage. Pediatr Res. 2012 Apr;71(4 Pt 2):474-81. doi: 10.1038/pr.2011.64. Epub 2012 Feb 8. PMID 22430383
- [Background] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Mesenchymal stem cell transplantation changes the gene expression profile of the neonatal ischemic brain. Brain Behav Immun. 2011 Oct;25(7):1342-8. doi: 10.1016/j.bbi.2011.03.021. Epub 2011 Apr 5. PMID 21473911
- [Background] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Nasal administration of stem cells: a promising novel route to treat neonatal ischemic brain damage. Pediatr Res. 2010 Nov;68(5):419-22. doi: 10.1203/PDR.0b013e3181f1c289. PMID 20639794
- [Background] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Repeated mesenchymal stem cell treatment after neonatal hypoxia-ischemia has distinct effects on formation and maturation of new neurons and oligodendrocytes leading to restoration of damage, corticospinal motor tract activity, and sensorimotor function. J Neurosci. 2010 Jul 14;30(28):9603-11. doi: 10.1523/JNEUROSCI.1835-10.2010. PMID 20631189
- [Background] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Mesenchymal stem cell treatment after neonatal hypoxic-ischemic brain injury improves behavioral outcome and induces neuronal and oligodendrocyte regeneration. Brain Behav Immun. 2010 Mar;24(3):387-93. doi: 10.1016/j.bbi.2009.10.017. Epub 2009 Oct 31. PMID 19883750
- [Background] van Velthoven CT, Kavelaars A, van Bel F, Heijnen CJ. Regeneration of the ischemic brain by engineered stem cells: fuelling endogenous repair processes. Brain Res Rev. 2009 Jun;61(1):1-13. doi: 10.1016/j.brainresrev.2009.03.003. Epub 2009 Apr 5. PMID 19348860
- [Background] Wagenaar N, Nijboer CH, van Bel F. Repair of neonatal brain injury: bringing stem cell-based therapy into clinical practice. Dev Med Child Neurol. 2017 Oct;59(10):997-1003. doi: 10.1111/dmcn.13528. Epub 2017 Aug 8. PMID 28786482
- [Background] Wagenaar N, de Theije CGM, de Vries LS, Groenendaal F, Benders MJNL, Nijboer CHA. Promoting neuroregeneration after perinatal arterial ischemic stroke: neurotrophic factors and mesenchymal stem cells. Pediatr Res. 2018 Jan;83(1-2):372-384. doi: 10.1038/pr.2017.243. Epub 2017 Nov 1. PMID 28949952
- [Derived] Wagenaar N, Baak LM, van der Aa NE, Groenendaal F, Dudink J, Tataranno ML, Koopman C, Verhage CH, Eijsermans RMJC, van Teeseling HC, Smit LS, Jellema RK, de Haan TR, Ter Horst HJ, de Boode WP, Steggerda SJ, Mulder-de Tollenaer SM, Dijkman KP, de Haar CG, de Vries LS, van Bel F, Heijnen CJ, Nijboer CH, Benders MJNL. Perinatal Arterial Stroke Treated With Stromal Cells Intranasally: 2-Year Safety and Neurodevelopment. Stroke. 2025 Sep;56(9):2410-2418. doi: 10.1161/STROKEAHA.125.050786. Epub 2025 Jul 14. PMID 40654084
- [Derived] Baak LM, Wagenaar N, van der Aa NE, Groenendaal F, Dudink J, Tataranno ML, Mahamuud U, Verhage CH, Eijsermans RMJC, Smit LS, Jellema RK, de Haan TR, Ter Horst HJ, de Boode WP, Steggerda SJ, Prins HJ, de Haar CG, de Vries LS, van Bel F, Heijnen CJ, Nijboer CH, Benders MJNL. Feasibility and safety of intranasally administered mesenchymal stromal cells after perinatal arterial ischaemic stroke in the Netherlands (PASSIoN): a first-in-human, open-label intervention study. Lancet Neurol. 2022 Jun;21(6):528-536. doi: 10.1016/S1474-4422(22)00117-X. PMID 35568047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Feb 11, 2020, and April 29, 2021,10 infants were included in the PASSIoN trial. Neonates were eligible for the study if they had been born at one of the ten neonatal intensive care units (NICU) in the Netherlands and had signs of suspected PAIS. All eligible patients were transferred to the NICU of the Wilhelmina Children's Hospital (part of the University Medical Center, Utrecht, Netherlands) for confirmation of PAIS by MRI, then MSC treatment, within 7 days after presentation.
Groups:
- Mesenchymal Stem Cells: Ten (near-)term newborns ≥36 weeks of gestation with or without clinical symptoms of PAIS but with a magnetic resonance imaging (MRI) confirmed PAIS (in the Middle Cerebral Artery region), and written parental consent were included this study.
  Mesenchymal Stem Cells: One dose of 50x10^6 bone marrow-derived allogeneic MSCs via the nasal route as soon as possible after confirmation of the stroke (in the middle cerebral artery), but within the first week of onset of presenting clinical symptoms. Within 30 minutes after cleaning the nose with saline, using standard procedures operative at the Neonatal Intensive Care Unit, the MSC will be delivered.
Period: Overall Study
Arm/Group | Mesenchymal Stem Cells
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mesenchymal Stem Cells
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: weeks of gestational age at birth] | 40.3 [39.9 to 41.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Birthweight [Median (Inter-Quartile Range); unit: gram] | 3415 [3140 to 3834]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Related to Intranasal MSC Treatment (Safety and Tolerability) in the Acute Setting.
Description: The primary objective is to determine if MSC treatment in neonates with PAIS is safe and tolerable in the acute setting. This will be measured by the number of Participants with treatment-related adverse events after MSC treatment.
Time Frame: 24 hours after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stem Cells
Number analyzed (Participants) | 10
Participants
  Serious adverse event: No | 10
  Serious adverse event: Yes | 0
  Adverse event: fever: No | 9
  Adverse event: fever: Yes | 1

2. Secondary Outcome: Number of Participants With Adverse Events Related to Intranasal MSC Treatment (Safety and Tolerability) in the Subacute/Long-term Setting
Description: The secondary objective is to determine subacute and long-term safety of MSC treatment at 3 months. This will be measured by the occurence of treatment-related adverse events after the initial hospital stay, such as infections or cerebral tumorigenicity on MRI. Follow-up assessment at 3 months is part of regular care for neonates with PAIS.
Time Frame: 3 months postnatal age
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stem Cells
Number analyzed (Participants) | 10
Participants
  no subacute adverse events until 3 months of age | 10
  subacute adverse events until 3 months of age | 0

ADVERSE EVENTS:
Time Frame: Treatment-related adverse events were monitored for 4 days after MSC administration (hospital stay), and until the age of 3 months (parent report).
Arm/Group | Mesenchymal Stem Cells
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mesenchymal Stem Cells (N=10)
Fever (General disorders) | 1 — One patient developed a fever of 38˚C 1 h after MSC administration that resolved spontaneously after 2 h, without clinical signs of distress or illness, and other vital parameters stayed within normal ranges.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT03356821/Prot_SAP_000.pdf